CLINICAL TRIAL: NCT03309683
Title: Clip Placement Following Colonic Endoscopic Mucosal Resection (EMR). The CLIPPER Study: A Nationwide Multi-center Randomized Clinical Trail
Brief Title: Clip Placement Following Colonic Endoscopic Mucosal Resection (EMR)
Acronym: CLIPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Maastricht University Medical Center (Other); Erasmus Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Maxima Medical Center (Other); Jeroen Bosch Ziekenhuis (Other); Bernhoven Hospital (Other); Isala (Other); Canisius-Wilhelmina Hospital (Other); Maasstad Hospital (Other); Noordwest Ziekenhuisgroep (Other); Meander Medisch Centrum (Other); Catharina Ziekenhuis Eindhoven (Other); Elisabeth-TweeSteden Ziekenhuis (Other); St Jansdal Hospital (Other); Leiden University Medical Center (Other); Dutch Digestive Diseases Foundation (Other); Franciscus Gasthuis (Other); Bravis Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R0003871
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2021-12

CONDITIONS: Polyp, Colonic; Bleeding
MeSH Terms: conditions — Colonic Polyps; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clip group (Experimental): Olympus Quick Clip Pro - Single Use Repositionable Clips will be used for Prophylactic clipping after EMR
  Interventions: Device: Olympus Quick Clip Pro - Single Use Repositionable Clips
- Control group (No Intervention): Standard treatment after EMR (as described in the detailed study description above)

INTERVENTIONS:
Device: Olympus Quick Clip Pro - Single Use Repositionable Clips — A hemoclip will be placed after every 0,5-1,0 cm of the resected area to proximate wound edges.
  Other Names: prophylactic clipping; hemoclip
  Arms: Clip group

SUMMARY:
Study design: A national, multi-center, patient-blinded, randomized clinical trial.

Study population: Patients undergoing EMR with a moderate to severe risk (right sided colon, ≥2cm) of developing Delayed Bleeding (DB).

Intervention: PC will be compared to standard care (no PC).

Main study endpoints: Primary endpoint is the incidence of DB. Secondary endpoints are cost-effectiveness, quality of life and (severe) adverse events related to PC, adenoma recurrence and risk factors for DB.

DETAILED DESCRIPTION:
Design

This is a multi-center, randomized, patient-blinded multicenter trial, comparing two treatment strategies in 356 patients undergoing EMR for a colonic lesion 2-6 cm. The study will be enrolled in a selection of academic and non-academic Dutch hospitals. Patients undergoing an EMR will be a randomly allocated by web-based randomization to:

A) PC treatment group: minimally 1 clip per 1 cm of the polyp resection plane: OR B) Control group: standard care: only clip placement in case of uncontrollable bleeding (not successfully managed by coagulation) AND/OR perforation.

Population The target population in this proposal includes patients of 18 years and older, who gave written informed consent, undergoing EMR of a colonic polyp with a moderate to severe risk of developing DB. Moderate-severe risk of DB is defined as a laterally spreading or sessile polyp morphology proximal to the splenic flexure, measuring 2-6cm. Given the significantly increased risk of bleeding in the cecum, ascending and transverse colon, clip placement at this location may have the greatest benefit.

Inclusion Gastroenterologists from participating hospitals of the Dutch EMR Study Group will be asked to recruit patients for the trial. They will provide written information about the trial to potential participants, i.e., all patients scheduled for an EMR of a (right-sided) colonic polyp 2-6 cm, and 18 years or older. Members of the study group will contact potentially eligible patients at the outpatient clinic, hospital wards or by phone and give detailed information about the trial. In- and exclusion criteria will be checked and questions about the trial will be answered. Eligible patients will be invited to participate. After both the patient and the study physician or nurse practitioner have signed the informed consent form, in- and exclusion criteria will be checked again and baseline measurements will be performed, which include disease specific questionnaires including risk-factors for DB (AC use, restarting AC, polyp size, visible vessel, etc) and generic and disease specific quality of life questionnaires (see below). Patient's contact details will be provided to the study center for randomization.

Standard of care (usual care) In Dutch common practice, PC is not standard of care. PC is used, based on the personal preference of the endoscopist, mostly in case of intra-procedural bleeding/(possible)perforation. In our study group the minority of endoscopists applies PC after EMR in case of high risk patients, defined as right-sided flat polyps of at least 2cm and on AC or AP therapy.

Definition clinical significant delayed bleeding (DB)

DB is defined as any bleeding occurring after the completion of the procedure necessitating blood transfusion, hospitalization, or re-intervention (either repeat endoscopy, angiography, or surgery). Self-limiting bleeding managed on an outpatient basis is not included. Severity of DB Severity of bleeding is defined according to the ASGE working party document for adverse events in colonoscopy:

1. Mild DB: any post-EMR medical consultation, unplanned hospital admission, or prolongation of hospital stays for 3 days or fewer.
2. Moderate DB: unplanned hospital admission of 4 to 10 days, transfusion, repeat endoscopy, any interventional radiology procedure, or intensive care unit (ICU) admission for 1 night.
3. Severe DB: admission to the ICU for more than 1 night, unplanned admission for more than 10 nights, surgery, or permanent disability.

Treatment of DB DB is primarily treated by resuscitation. In case of resuscitation failure, colonoscopy, angiography with coiling and eventually surgery may be applied to control the bleeding site.

Follow-up After the EMR patients are contacted at 30, 90 and 180 days (short-term and long-term effects). At 180 days a colonoscopy is scheduled to access the adenoma recurrence rate (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* laterally spreading or sessile polyp morphology (Paris classification 0-IIa/b/c) proximal to the splenic flexure, measuring 2-6 cm
* All patients aged >18 years undergoing an EMR
* Written informed consent

Exclusion Criteria:

* Previous resection or attempted resection of a lesion less than 30 days ago or in the same session,
* Clip deployed prior to the completion of the EMR for a perforation or a major intra-procedural bleeding not treatable by coagulation,
* Endoscopic appearance of invasive malignancy (non-lifting Kato D, Kudo V pit pattern),
* Pregnancy,
* Active inflammatory colonic conditions (e.g. inflammatory bowel disease),
* Insufficiently corrected anticoagulants AND/OR a clotting disorder (platelet count <50x109/l, INR > 1,5),
* American Society of Anesthesiology (ASA) Grade IV-V,
* Macroscopic non-radical resection,
* >1 lesion in 1 session,
* Involvement of valvula Bauhin or appendiceal orificium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Delayed bleeding | 30 days
  Clinical relevant delayed bleeding defined according to the ASGE working party document for adverse events in coloscopy.

SECONDARY OUTCOMES:
Adenoma recurrence | 180 days
  Recurrence rate will be determined by endoscopy and biopsies.
Cost-effectiveness | 180 days
  A cost effectiveness analysis will be done, based on length of hospital stay and professional medical attendance and aided by an estimation of the impact on quality of health by the questionnaires EQ-5D, iMCQ, iPCQ.
EMR scar evaluation | 180 days
  EMR scars will be evaluated by endoscopic photography and biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Erwin JM Van Geenen, dr, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Ziekenhuis St Jansdal, Harderwijk, Gelderland
  - Radboudumc, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: No
Open for sharing IPD after study completion and publication. Currently not yet applicable as the study is still recruiting.

REFERENCES:
- [Derived] Kemper G, Turan AS, Schreuder RM, Schrauwen RWM, Hadithi M, Didden P, Bastiaansen BAJ, van der Spek BW, Droste JSTS, Schwartz MP, Hazen WL, Straathof JWA, Boonstra JJ, Alkhalaf A, Voogd FJ, Allajar D, de Graaf W, Koehestanie P, Roomer R, de Ridder RJJ, Moons LMG, Siersema PD, van Geenen EJM; Dutch EMR Study Group. The effect of prophylactic clipping on delayed bleeding after proximal colonic endoscopic mucosal resection: a multicenter, randomized controlled trial (CLIPPER). Endoscopy. 2025 Nov;57(11):1243-1250. doi: 10.1055/a-2637-3180. Epub 2025 Jul 22. PMID 40695477
- [Derived] Turan AS, Moons LMG, Schreuder RM, Schoon EJ, Terhaar Sive Droste JS, Schrauwen RWM, Straathof JW, Bastiaansen BAJ, Schwartz MP, Hazen WL, Alkhalaf A, Allajar D, Hadithi M, van der Spek BW, Heine DGDN, Tan ACITL, de Graaf W, Boonstra JJ, Voogd FJ, Roomer R, de Ridder RJJ, Kievit W, Siersema PD, Didden P, van Geenen EJM; Dutch EMR Study Group. Clip placement to prevent delayed bleeding after colonic endoscopic mucosal resection (CLIPPER): study protocol for a randomized controlled trial. Trials. 2021 Jan 18;22(1):63. doi: 10.1186/s13063-020-04996-7. PMID 33461579